CLINICAL TRIAL: NCT01699438
Title: Mesalazine Treatment in IBS, a Double-blind Placebo-controlled Phase II Intervention Study in Adult Patients
Brief Title: Mesalazine Treatment in IBS (The MIBS Study)
Acronym: MIBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hans Törnblom (Other)
Collaborators: Sahlgrenska University Hospital (Other); Smerud Medical Research International AS (Other); Alimenta AB (Unknown); Tillotts Pharma AG (Industry); Karolinska University Hospital (Other); Haukeland University Hospital (Other); Oslo University Hospital (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor-Investigator, Hans Törnblom, MD, PhD, Göteborg University
Organization: Göteborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-2268
Record Dates: First submitted 2012-09-16; First posted 2012-10-03 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Inflammation; Mesalazine
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesalazine (Experimental)
  Interventions: Drug: Mesalazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalazine — 2400 mg q.d. for 8 weeks
  Other Names: Asacol
  Arms: Mesalazine
Drug: Placebo — 3 tablets q.d. for 8 weeks
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a condition characterised by abdominal pain or discomfort in combination with altered bowel function (stool frequency and/or stool consistency), currently defined by the Rome III criteria. The current IBS definition specifies that there are no structural or biochemical abnormalities to account for the symptoms but there is growing evidence that in at least a subset of IBS patients, a discrete immune activation might be a key pathogenetic factor. The condition is prone to develop after a gastroenteritis, post-infectious IBS, and increased numbers of lymphocytes, mast cells and pro-inflammatory cytokines like Interleukin (IL)-1β, IL-6, Tumor necrosis factor (TNF)-α and a general increase in mucosal cellularity have been reported. Despite this, the efficacy of anti-inflammatory agents has been poorly investigated.

This will be a randomised, double blind, placebo-controlled, parallel-group, multi-centre study that aims to include a total of 200 subjects with irritable bowel syndrome (IBS). All subjects will be randomised to receive either 3x800 mg of mesalazine (Asacol®) or corresponding placebo once daily for a total treatment duration of 8 weeks. Males and females aged 18 to 70 years who already are diagnosed with IBS based on the Rome III diagnostic criteria and with a symptom intensity of at least moderate level; defined as an IBS Severity Scoring System (IBS-SSS) score of ≥175 at both Screening (Visit 1, Day -21±2) and Baseline (Visit 2, Day 0) will be eligible to enter the study.

Primary aim:

To assess the effect of mesalazine (Asacol®) treatment compared to placebo on global IBS symptoms: A treatment responder will be defined by answering the satisfactory relief of IBS-symptoms question "yes" at the end of at least 4 out of of 8 treatment weeks.

Secondary aims:

To assess mesalazine (Asacol®) treatment compared to placebo regarding:

1. Levels of inflammatory mediators in the rectal mucosa (e.g. neutrophil mediators, eosinophilic mediators, mast cell activity mediators and cytokines) measured by a new diagnostic tool, the Mucosal Patch Technology (MPT) by means of Enzyme-Linked Immunosorbent Assays (ELISA)
2. Effects on number of immune cells (count per high power field) and cytokine content (immunohistochemistry) in mucosal biopsies
3. Calprotectin levels in faeces (mg/kg)
4. Individual IBS symptom parameters derived from a symptom diary and also measured by IBS-SSS

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 70 years, both inclusive
* Subject is diagnosed with irritable bowel syndrome (IBS) prior to Screening based on the Rome III diagnostic criteria.
* Subject presents with IBS symptom intensity of at least moderate level; defined as an IBS Severity Scoring System (IBS-SSS) score of ≥175 at both Screening (Visit 1, Day -21±2) and Baseline (Visit 2, Day 0)
* Provision of signed informed consent

Exclusion Criteria:

* Subjects who are unable to understand the written and verbal instructions
* Presence of a systemic inflammatory disease
* Presence of other gastrointestinal diseases likely to explain the IBS symptoms
* Presence of other severe somatic disease
* Treatment with non-steroidal anti-inflammatory drugs (NSAID), opioid analgetics or acetylsalicylic acid (ASA) compounds within 7 days prior to screening (Visit 1, Day -21±2)
* Treatment with systemic antibiotics within 28 days prior to Screening (Visit 1, Day -21±2)
* Treatment with immunosuppressant drugs within 28 days prior to Screening (Visit 1, Day -21±2)
* Other significant medical treatment, which, in the opinion of the investigator, may compromise the safety and efficacy objectives of the study, within 28 days prior to Screening (Visit 1, Day -21±2)
* Previously confirmed allergy towards ASA or mesalazine
* Presence of renal disease and/or concomitant treatment with medications with potential renal side effects
* Current ongoing infection
* History of, or current, drug or alcohol dependence
* Pregnant or lactating women
* Subjects suspected not to follow instructions based on the discretion of the Investigator
* Current participation in other intervention studies
* Female subjects of childbearing potential unwilling to use adequate contraceptive measures throughout the duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Global Irritable Bowel Syndrome (IBS) symptoms | 8 weeks
  The main measurement parameter of symptom alleviation will be a weekly question regarding satisfactory relief of global IBS symptoms. A treatment responder will be defined as answering "yes" ≥50% of the weeks (≥4 weeks)

SECONDARY OUTCOMES:
Inflammatory mediators | 8 weeks
  Measured by the Mucosal Patch Technology (MPT), e.g. neutrophil mediators (myeloperoxidase (MPO)), eosinophilic mediators (eosinophil cationic protein (ECP)), mast cell activity mediators (tryptase) and cytokines (Interleukin (IL)-2, IL-6, Tumor necrosis factor (TNF)-alpha, IL-1beta etc) by Enzyme-Linked Immunosorbent Assays (ELISA), (ug/ml).
Effect on immune cells and cytokines in mucosal biopsies | 8 weeks
  Counts per high-power field in microscopy and by immunohistochemistry
Levels of calprotectin in faeces | 8 weeks
  Enzyme-Linked Immunosorbent Assay (ELISA), mg/kg
Change in total IBS symptom severity score (IBS-SSS) | 8 weeks
  Absolute change in IBS-SSS compared to baseline.
Individual symptom parameters in IBS symptom severity score (IBS-SSS) and the IBS diary | 8 weeks
  Reduction of scores regarding individual question components (visual analog scale (VAS)) in IBS-SSS. Stool frequency and consistency expressed by Bristol Stool Form Scale in a separate IBS diary.
Exploratory responder variables | 8 weeks
  1. Satisfactory symptom relief ≥75% of the time
  2. Reduction in IBS-SSS ≥50 at end of treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hans Törnblom, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Huddinge
  - Norrland's University Hospital, Umeå